CLINICAL TRIAL: NCT05164887
Title: Can we Manipulate the Bowel Microbiota and Prevent Anastomotic Leakage in Colorectal Laparoscopic Surgery? Preliminary Results of the MIRACLe Study.
Brief Title: Microbiota Implementation to Reduce Anastomotic Colorectal Leaks (MIRACLe)
Acronym: MIRACLe
Status: Completed | Type: Observational
Sponsor: S.Eugenio Hospital (Other)
Collaborators: Domenico Spoletini, M.D. PhD (Unknown); Michele Grieco, M.D. (Unknown); Rosa Marcellinaro, M.D PhD (Unknown); Andrea Mingoli, M.D. PhD (Unknown); Rosa Menditto, M.D. (Unknown); Vincenzo Napoleone, PhD (Unknown); Gioia Brachini, M.D. PhD (Unknown)
Responsible Party: Principal Investigator, Massimo Carlini, Head of Department of Surgery - Head of General Surgery Unit, S.Eugenio Hospital
Other Study IDs: 1.0
Record Dates: First submitted 2021-12-03; First posted 2021-12-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Surgery; LAP; Anastomotic Leak; Microbial Substitution
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- MIRACLe patients: Patient affected by colorectal cancer submitted to laparoscopic resection with MBP + OA + perioperative Probiotics administration.
  MBP = oral polyphosphate 500ml preoperative OA = Amoxicillin/Clavulanic acid 1g x 2 + metronidazole 250mg x 3 Probiotics = Streptococcus thermophilus; Bifidobacterium breve; Bifidobacterium longum; Bifidobacterium infantis; Lactobacillus acidophilus; Lactobacillus plantarum; Lactobacillus paracasei; Lactobacillus delbrueckii subsp. Bulgaricus 4,4g x 2
  Interventions: Procedure: Laparoscopic colorectal resection

INTERVENTIONS:
Procedure: Laparoscopic colorectal resection — the patients candidate to laparoscopic colorectal resection for cancer are perioperatively treated with mechanical bowel preparation, oral antibiotics and administration of probiotics
  Other Names: Perioperative bowel preparation

SUMMARY:
Aim of this study is to implement the intestinal microbiota by perioperative administration of probiotics, oral antibiotics and low volume mechanical preparation in order to reduce the incidence of colorectal anastomotic leaks and dehiscences.

DETAILED DESCRIPTION:
Anastomotic leaks and dehiscences are still the most frequent complication of colorectal surgery and have a multifactorial etiology.

Microbiota refers to the totality of microorganisms in a defined environment. The Microbiome represents the set of genomes of all microorganisms and its environmental relationships. The microbiome performs various and important functions, but above all it contributes to maintaining the integrity of the mucous barrier of the intestinal epithelium.

The composition, biodiversity and functions of the intestinal microbiota vary both longitudinally along the entire intestinal tract from the mouth to the anus, and radially from the muco-epithelial layer to the intestinal lumen. This biodiversity fluctuates with daily variations following various conditions such as diet, physical activity, interactions with people and animals, etc., but remains stable in healthy subjects.

Particular conditions can determine a phenotypic shift of some bacterial families with the development of species with different characteristics, potentially pathogenic which can favor the onset of fistulas and anastomotic dehiscences in experimental setting.

It is known experimentally that the surgical act alone causes a greater change in the composition of the intestinal microbiota. The way in which surgical stress alters the microbiome lies in the mechanisms which the host and the microorganisms communicate. It has recently been shown that mechanical bowel preparation and the administration of antibiotics have an influence on the microbiome. In particular, the mechanical preparation with polyethylene glycol (PEG) and oral antibiotics (OA) can constitute a positive element for surgical outcomes, while intravenous antibiotics very often affect microbiota negatively.

The intestinal flora influence the healing of intestinal anastomoses and non-pathogenic saprophytes allow anastomoses to withstand increased endoluminal pressures. Based on this, it has been shown that the postoperative implementation of bifidobacteria improves functional recovery, reduces the inflammatory response and improves the composition of the fecal microbiota in patients undergoing colorectal surgery.

Based on these considerations, this study aims to modify the preoperative preparation by implementing the intestinal microbiota in order to evaluate the incidence of anastomotic leaks.

The patient's treatment will be divided into 3 phases: preoperative, intraoperative and postoperative.

Preoperative treatment The preoperative phase runs from the fifth preoperative day (-5) to day -1.

In this phase, patients will undergo microbiota implementation through preoperative preparation consisting of:

* Oral probiotics: Streptococcus thermophilus; Bifidobacterium brevis; Bifidobacterium longum; Bifidobacterium infantis; Lactobacillus acidophilus; Lactobacillus plantarum; Lactobacillus paracasei; Lactobacillus delbrueckii subsp. Bulgaricus (VSL # 3) 4,4gr, equal to 450 billion live bacterial cells, every 12 hours from the day -5.
* Oral antibiotic prophylaxis with Amoxicillin / Ac. Clavulanic (Augmentin), 1g every 12 hours + Metronidazole (Flagyl), 250 mg every 8 hours in the day -1.
* Mechanical preparation with Polyethylene Glycol - low volume.

Intraoperative treatment - Surgical technique Under general anesthesia and hemodynamic monitoring, pneumoperitoneum induction and positioning of the trocars necessary for the execution of the surgery will be carried out. The number and location of the trocars will be determined by the type of intervention to be performed and the operator's preferences. After an abdominal exploration, we will continue with the resective phase of the intervention depending on the location of the disease and in compliance with the oncological radicality criteria. The anastomosis will be performed according to the principles of good vascularization and reconstruction without tension or torsion.

The anastomosis will be:

* Intracorporeal (mechanical / manual) if ileo-colic.
* Intra- or extra-corporeal (mechanical or manual respectively) if colocolic, after resection of the transverse, splenic or segmental flexure of the left colon.
* Transanal (mechanical) if colorectal, after left hemicolectomy, sigmoidectomy or resection of the rectum (both intra- and subperitoneal).

The positioning of nasogastric tube, drains, bladder catheter, central vascular accesses, whose management will be at the discretion of the operators, is subject to the Enhanced Recovery After Surgery (ERAS®) principles in use in the centers participating in the study.

- Intraoperative phase On the morning of the surgery, antibiotics will be administered: Amoxicillin / Ac. Clavulanic 1g + Metronidazole 250 mg orally, about 2 hours before the induction of anesthesia.

Anastomotic endoluminal instillation of a dose (4.4 g) of the probiotic used in the preoperative phase, diluted in 20cc of sterile physiological solution, will also be performed. This dose will be equally distributed in the 2 intestinal stumps. The instillation will take place using a special laparoscopic cannula.

Postoperative treatment The postoperative management of patients will be based on compliance with Enhanced Recovery After Surgery (ERAS®) principles, where applicable (nasogastric tube removal on first postoperative day, bladder catheter removal on first postoperative day, early feeding, mobilization, etc.).

The oral antibiotic prophylaxis will be continued until day +1, while the administration of probiotics will take place until day +4.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ASA I - II - III
* Colorectal cancer
* Elective surgery
* Laparoscopic resections

Exclusion Criteria:

* Age < 18 years
* ASA IV
* Emergency surgery
* Laparotomic resections
* Diverticular disease or IBD
* Hartmann or Miles procedures
* Stomies
* Major intraoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by colorectal cancer submitted to laparoscopic resections with ileo- colo- rectal anastomoses
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Fistulas and Anastomotic Leaks | 4 weeks
  Evaluation of incidence of AL compared to a group of 500 colorectal resection in patient prepared with ev antibiotics, no MBP and without probiotics administration

SECONDARY OUTCOMES:
Incidence of SSI | 4 weeks
  Measuring incidence of surgical site infections compared to the control group

CONTACTS AND LOCATIONS:
Locations (1):
- S Eugenio Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No